CLINICAL TRIAL: NCT04310930
Title: Finding the Optimal Regimen for Mycobacterium Abscessus Treatment (FORMaT)
Brief Title: Finding the Optimal Regimen for Mycobacterium Abscessus Treatment
Acronym: FORMaT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Australian Government Department of Health and Ageing (Other Government); Children's Hospital Foundation (Other); Cystic Fibrosis Foundation (Other); Newcastle University (Other); Griffith University (Other); Erasmus Medical Center (Other); Monash University (Other); University of Copenhagen (Other); South Australian Health and Medical Research Institute (Other); University of Melbourne (Other); Murdoch Childrens Research Institute (Other); QIMR Berghofer Medical Research Institute (Other)
Responsible Party: Principal Investigator, Claire Wainright, Professor, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1209-0672
Record Dates: First submitted 2020-02-28; First posted 2020-03-17 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Disease Due to Mycobacteria (Diagnosis)
Keywords: Mycobacterium abscessus; Pulmonary disease; Microbiological; Regimen; Radiological; Quality of life; Health economics; Biomarkers
MeSH Terms: conditions — Disease; Mycobacterium Infections, Nontuberculous; Lung Diseases | interventions — Amikacin; Tigecycline; Imipenem; Cefoxitin; Azithromycin; Clarithromycin; Clofazimine; Ethambutol; Linezolid; Trimethoprim, Sulfamethoxazole Drug Combination; Doxycycline; Moxifloxacin; bedaquiline; Rifabutin

STUDY DESIGN:
Intervention Model Description: There are 2 different phases of treatment; intensive therapy (IT) followed by consolidation therapy (CT). Intervention cohort participants will be randomised to 1 of 3 treatment arms for 6 weeks of IT. After the first 6 weeks of IT participants who are culture positive for MABS are randomised to either prolonged IT (additional 6 weeks of IT) then CT, or to commence CT. If, at week 6 participants are MABS culture-negative they will commence CT. Participants commencing CT are randomised to one of two treatment arms for 50 weeks. There are 12 possible paths through the trial. This standing platform trial design enables assessment of short IT, prolonged IT, and CT components individually as well as the overall combination of IT and CT. After 100 patients have completed short IT an interim analysis will be conducted, and Bayesian adaptive randomisation (BAR) will be implemented. New interventions may be added or stopped in the future due to lack of benefit at interim analyses.
Masking Description: The FORMAT trial may include placebo controlled double blind randomised interventions in the future, but the initial intervention program is randomised but open label.
  There will be three stages of randomisation in the intervention program of this study, dictating the treatment the participant will receive. Randomisation at each level will be conducted using the method of minimisation. Each randomisation level will be planned to enable flexibility via pre-planned adaptations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Intensive Therapy A (Active Comparator): Following Randomisation 1, Participants will receive intensive drug therapy in the form of IV amikacin, IV tigecycline, IV cefoxitin/imipenem + oral azithromycin AND clofazimine.
  Interventions: Drug: Amikacin; Drug: Tigecycline; Drug: Imipenem; Drug: Cefoxitin; Drug: Azithromycin; Drug: Clarithromycin; Drug: Clofazimine; Drug: Ethambutol
- Intensive Therapy B (Experimental): Following Randomisation 1, Participants will receive inhaled amikacin (IA), IV tigecycline, IV cefoxitin/imipenem + oral azithromycin/oral clarithromycin AND clofazimine.
  Interventions: Drug: Tigecycline; Drug: Imipenem; Drug: Cefoxitin; Drug: Azithromycin; Drug: Clarithromycin; Drug: Clofazimine; Drug: Ethambutol; Drug: Amikacin
- Intensive Therapy C (Experimental): Following Randomisation 1, Participants will receive intensive drug therapy in the form of IV amikacin, IV tigecycline, IV cefoxitin/imipenem + oral azithromycin/oral clarithromycin.
  Interventions: Drug: Amikacin; Drug: Tigecycline; Drug: Imipenem; Drug: Cefoxitin; Drug: Azithromycin; Drug: Clarithromycin; Drug: Ethambutol
- Consolidation A (Active Comparator): Oral clofazimine + oral azithromycin/oral clarithromycin in combination with one to three of the following oral antibiotics: oral linezolid, oral co-trimoxazole, oral doxycycline, oral moxifloxacin, oral bedaquiline (adults only), oral rifabutin.
  Interventions: Drug: Azithromycin; Drug: Clarithromycin; Drug: Clofazimine; Drug: Ethambutol; Drug: Linezolid; Drug: co-trimoxazole; Drug: Doxycycline; Drug: Moxifloxacin; Drug: Bedaquiline; Drug: Rifabutin
- Consolidation B (Experimental): Inhaled amikacin (IA), oral clofazimine + oral azithromycin/oral clarithromycin in combination with one to three of the following oral antibiotics: oral linezolid, oral co-trimoxazole, oral doxycycline, oral moxifloxacin, oral bedaquiline (adults only), oral rifabutin.
  Interventions: Drug: Azithromycin; Drug: Clarithromycin; Drug: Clofazimine; Drug: Ethambutol; Drug: Amikacin; Drug: Linezolid; Drug: co-trimoxazole; Drug: Doxycycline; Drug: Moxifloxacin; Drug: Bedaquiline; Drug: Rifabutin

INTERVENTIONS:
Drug: Amikacin — Adults: Intravenous amikacin 5mg/kg once daily or 7.5mg/kg twice daily or 20-25 mg/kg thrice weekly. Children:Intravenous amikacin 15-30 mg/kg once daily, maximum dose 1500mg
  Arms: Intensive Therapy A; Intensive Therapy C
Drug: Tigecycline — Adults: Intravenous Tigecycline 25 mg increasing by 5 mg every two doses until either maximum dose reached (50mg) or until patient is unable to tolerate twice daily. Children (≥8 years of age) intravenous tigecycline: Day 1- 0.6mg/kg twice daily to a maximum of 25mg. Day 2- 0.6mg/kg (maximum 25mg) in the morning, 1.2 mg/kg (maximum 50mg) at night. Day 3- 1.2mg/kg (maximum 50 mg) twice daily
  Arms: Intensive Therapy A; Intensive Therapy B; Intensive Therapy C
Drug: Imipenem — Adults: Intravenous Imipenem (≥50kg) 500mg twice daily (<50kg) 15 mg/kg twice daily. Children: intravenous imipenem Day 1- 2- 25mg/kg (maximum 1g) twice daily. DAY 3- 25mg/kg (maximum 1g) four times daily (drop to 3 if not tolerated).
  Arms: Intensive Therapy A; Intensive Therapy B; Intensive Therapy C
Drug: Cefoxitin — Adults: If imipenem is poorly tolerated intravenous cefoxitin 200 mg/kg thrice daily. Children: if imipenem is poorly tolerated intravenous cefoxitin 50mg/kg (maximum 4g) four times daily.
  Arms: Intensive Therapy A; Intensive Therapy B; Intensive Therapy C
Drug: Azithromycin — Adults: Oral azithromycin 500mg (≥40kg) once daily, (<40kg) 250mg once daily.During consolidaiton: 500mg (≥40kg) thrice weekly, (<40kg) 250mg thrice weekly.
  Children: Oral azithromycin:10mg/kg (maximum 500mg) once daily. During consolidation 10mg/kg once daily maximum 500mg.
Drug: Clarithromycin — Adult: If azithromycin is poorly tolerated use oral clarithromycin 500mg twice daily.Children: If azithromycin is poorly tolerated use oral clarithromycin. In children 1 month old- 11years of age the following dosing applies: <8kg: 7.5mg/kg twice daily, maximum dose 62.5mg, 8-11kg: 62.5mg twice daily, maximum dose 62.5mg, 12-19 kg: 125mg twice daily, maximum dose 125mg, 20-29 kg: 187.5mg twice daily, maximum dose 187.5mg, 30-40 kg: 250mg twice daily, maximum dose 250mg, Children 12-18 years of age: 500 mg twice daily
Drug: Clofazimine — Adult: Oral clofazimine 100mg once daily. Children: Oral clofazimine: 3-5mg/kg once daily. Maximum dose of 50mg once daily if <40kg or 100mg if ≥40kg once daily.
  Arms: Consolidation A; Consolidation B; Intensive Therapy A; Intensive Therapy B
Drug: Ethambutol — Adults: with confirmed mixed NTM infections (slow growers + MABS) oral ethambutol can be added at either 15 mg/kg once daily or 25mg/kg thrice weekly. Children with confirmed mixed NTM infections (slow growers + MABS) oral ethambutol can be added at 20 mg/kg once daily.
Drug: Amikacin — adult: Inhaled amikacin 500mg twice daily. Children: Inhaled amikacin 500mg twice daily
  Arms: Consolidation B; Intensive Therapy B
Drug: Linezolid — Adult: during consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin, bedaquiline or rifabutin) guided by participant susceptibility and tolerance. Oral linezolid 600mg once daily.
  Children: during consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin or rifabutin) guided by participant susceptibility and tolerance. Age 1 week - 9 years 10mg/kg twice daily maximum dose of 300mg. Age 10-12 years 10mg/kg twice daily maximum dose of 600mg. >12 years 600mg once daily.
  Arms: Consolidation A; Consolidation B
Drug: co-trimoxazole — Adult: during consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin, bedaquiline or rifabutin) guided by participant susceptibility and tolerance. Oral Co-trimoxazole (TMP-SMX) 160/800mg twice daily. Children: During consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin or rifabutin) guided by participant susceptibility and tolerance. Oral co-trimoxazole 5mg TMP/kg maximum dose of 160mg TMP/ 800mg SMX twice daily.
  Arms: Consolidation A; Consolidation B
Drug: Doxycycline — Adult: during consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin, bedaquiline or rifabutin) guided by participant susceptibility and tolerance. Oral doxycycline 100mg once daily. Children: During consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin or rifabutin) guided by participant susceptibility and tolerance. Oral doxycycline (ages ≥ 8 years) 2mg/kg once daily maximum dose 100mg.
  Arms: Consolidation A; Consolidation B
Drug: Moxifloxacin — Adult: during consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin, bedaquiline or rifabutin) guided by participant susceptibility and tolerance. Oral moxifloxacin 400mg once daily. Children: During consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin or rifabutin) guided by participant susceptibility and tolerance. Oral moxifloxacin 10-15mg/kg once daily, maximum dose 400mg
  Arms: Consolidation A; Consolidation B
Drug: Bedaquiline — Adult: during consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin, bedaquiline or rifabutin) guided by participant susceptibility and tolerance. Oral bedaquiline (18-64 years of age) 400mg once daily for the first two weeks followed by 400mg thrice weekly for 22 weeks (maximum duration of 6 months).
  Arms: Consolidation A; Consolidation B
Drug: Rifabutin — Adult: during consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin, bedaquiline or rifabutin) guided by participant susceptibility and tolerance. Oral rifabutin: 5mg/kg once daily, maximum 300-450mg. Children: During consolidation in combination with one to three oral antibiotics (co-trimoxazole, doxycycline, moxifloxacin or rifabutin) guided by participant susceptibility and tolerance. Oral rifabutin 5mg/kg once daily
  Arms: Consolidation A; Consolidation B

SUMMARY:
Mycobacterium abscessus (MABS) is a group of rapid-growing, multi-drug resistant non-tuberculous mycobacteria (NTM) causing infections in humans. MABS pulmonary disease (MABS-PD) can result in significant morbidity, increased healthcare utilisation, accelerated lung function decline, impaired quality of life, more challenging lung transplantation, and increased mortality. While the overall numbers affected is small, the prevalence of infections is increasing worldwide. The Finding the Optimal Regimen for Mycobacterium abscessus Treatment (FORMaT) trial aims to produce high quality evidence for the best treatment regimens to maximise health outcomes and minimise toxicity and treatment burden, as well as developing biomarkers (serology, gene expression signatures, and radiology) to guide decisions for starting treatment and measuring disease severity in patients with MABS PD.

DETAILED DESCRIPTION:
Mycobacterium abscessus (MABS) are a group of non-tuberculous mycobacteria (NTM) found in water and soil habitats that exhibit high levels of intrinsic multi-drug resistance. They are recognised opportunistic human pathogens capable of causing chronic pulmonary disease (MABS-PD), predominantly in individuals with underlying inflammatory lung diseases.

Finding the Optimal Regimen for Mycobacterium abscessus Treatment (FORMaT) is an iterative, standing, platform trial with innovative and adaptive properties that evaluate and develop the optimal combinations of therapies for children and adults with MABS-PD to clear MABS infection with acceptable tolerance. We will use these opportunities afforded by the clinical trial platform to establish discovery studies to: (i) understand the effects of disease and treatment on health-related quality of life, (ii) determine cost effectiveness of interventions, (iii) optimise pharmacokinetic drug dosing, (iv) understand susceptibility to MABs-PD, (v) develop biomarkers of clinical disease, (vi) investigate genomics of MABs strains causing MABs-PD and development of antimicrobial resistance.

FORMaT provides a pragmatic design to address challenges to develop an evidence base for the first time for MABS-PD. Initially, the trial has been designed to test therapies that are currently the basis for treatment guidelines for MABS-PD. The trial has the capacity to add new treatments and to eliminate therapies because of futility as they either lack efficacy or cause unacceptable toxicity. Novel therapeutic approaches are then tested against the previously determined optimal approaches, thus leading in an iterative fashion to improve microbiological clearance, and health outcomes associated with MABS-PD. The trial is designed as a series of trials within the main trial to enable investigation of the different phases of treatment; intensive (intravenous treatment phase) and consolidation (oral and or inhaled treatment phase) based on clinical guidelines. The primary outcome for each trial is microbiological clearance with clinical tolerance (Grade 1 or 2) based on Common Terminology Criteria for Adverse Events (version 5). This enables subjects to continue in the trial even if tolerance is poor or they change treatments in a specific phase of the trial as those events contribute to the primary outcome determination.

ELIGIBILITY:
Eligibility criteria for the FORMaT trial can be applied at two levels:

1. Eligibility into the Intervention Program, or;
2. Eligibility into the Observational Cohort.

Potential participants can only be enrolled in either the Intervention Program or the Observational Cohort at any one time. Provided the eligibility criteria are met, potential participants may either:

1. Enrol directly into the Intervention Program, or;
2. Enrol into the Observational Cohort and transition into the Intervention Program once they satisfy the inclusion criteria for this program which can occur at any time during the trial.

Eligibility into the FORMaT trial will be assessed at screening. Observational Cohort participants who go on to meet the Intervention Program eligibility criteria can transition from the Observational Cohort to the Intervention Program.

INTERVENTION PROGRAM ELIGIBILITY (APPENDIX A) Potential participants are eligible for the Intervention Program (Appendix A) if the criteria below are met. Eligible participants with mixed NTM infections (slow growers + MABS) or with recurrence of MABS infection following completion of previous treatment will be eligible if they meet the inclusion and exclusion criteria listed below. For eligible participants with mixed NTM infections additional therapy combinations are available as detailed in the relevant appendices.

INTERVENTION PROGRAM INCLUSION CRITERIA

1. Positive MABS-PD diagnosis meeting all three American Thoracic Society clinical, radiological and microbiological diagnostic criteria for MABS-PD. Defined as:

   1. Clinical: Pulmonary symptoms and exclusion of other diagnoses.
   2. Radiological: Nodular or cavitary opacities on chest radiograph or a chest high-resolution computed tomography (HRCT) scan showing multifocal bronchiectasis with multiple small nodules.
   3. Microbiological: MABS positive culture results from at least two separate expectorated sputum samples.

   or Positive culture results from at least one bronchial wash or lavage. or Transbronchial or other lung biopsy with mycobacterial histopathologic features (granulomatous inflammation or acid-fast bacilli (AFB)) and positive culture for NTM or biopsy showing mycobacterial histopathologic features (granulomatous inflammation or AFB) and one or more sputum or bronchial washes that are culture positive for NTM.

   Screening samples must be collected within the timeframes stated in the relevant appendix.
2. Male or female participants of any age.
3. Participant has not received treatment for MABS-PD in the 12 months preceding assessment of eligibility or as specified in the relevant appendix (this includes drugs prescribed for the treatment of other mycobacteria and/or other indications that may have activity against MABS, as specified in the FORMaT Prohibited Drug List Standard Operating Procedure (SOP)).
4. Informed consent signed by participant or parent/legal guardian if participant is under 18 years of age.
5. Ability to comply with study visits, therapies and study procedures as judged by the site investigator.

INTERVENTION PROGRAM EXCLUSION CRITERIA

* Participants receiving current treatment for MABS (this includes drugs prescribed for the treatment of other mycobacteria and/or other indications that may have activity against MABS, as specified in the FORMaT Prohibited Drug List SOP), except for participants taking azithromycin as part of routine treatment for CF or chronic infection-related pulmonary disease, or as specified in the relevant appendix.
* Participants who have a QTc interval of >500 milliseconds (QT interval corrected based on Fridericia method).
* Participants who are pregnant or planning to continue breast feeding.
* Known hypersensitivity or contraindication to any of the therapies for which no alternative option(s) have been provided.

OBSERVATIONAL COHORT INCLUSION CRITERIA

To be eligible to participate in the Observational Cohort the following criteria must be met:

1. Male and female participants of any age with at least one positive respiratory culture for MABS.
2. Informed consent signed by participant or parent/legal guardian if participant is under 18 years of age.
3. Ability to comply with study visits and study procedures as judged by the site investigator.

OBSERVATIONAL COHORT EXCLUSION CRITERIA

Potential participants will be ineligible to participate in the Observational Cohort if any of the following criterion are met:

• Receiving active treatment for MABS within the previous 12 months (this includes drugs prescribed for the treatment of other mycobacteria and/or other indications that may have activity against MABS, as specified in the FORMaT Prohibited Drug List SOP, except for participants taking azithromycin as part of routine treatment for CF or chronic infection-related pulmonary disease).

ADDITIONAL ELIGIBILITY CRITERIA Mixed NTM infections Participants who have cultured slow growing NTM of the same species two or more times in the 24 months prior to screening, with one of those cultures within the 6 months prior to screening, will be considered to have mixed NTM infection at the time of screening. The participants must meet all other inclusion criteria and no exclusion criteria to be eligible for participation. Ethambutol may be used in addition to trial therapies to cover mixed NTM infections considered to require treatment by their clinician.

Appendix specific sub-studies and integrated studies Appendix specific sub-studies and integrated studies may have additional eligibility criteria which are described in each of the relevant appendices.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the Intervention Program is microbiological clearance of MABS with good tolerance of the interventions. | Screening (Day 0) to End of treatment plus four weeks off-treatment (Final Outcome Visit (Week 56 for those allocated to Immediate Consolidation or Week 62 for those allocated to Prolonged Intensive).
  The primary outcome of the Intervention Program is microbiological clearance of MABS with good tolerance of the interventions.
  Definition of MABS clearance at final outcome:
  Negative MABS cultures from four consecutive sputum samples with one of those sputum specimens collected four weeks after the completion of consolidation therapy, or a MABS negative Bronchoalveolar Lavage (BAL) collected four weeks after completion of consolidation.
  Definition of tolerance:
  Tolerance is based on the Common Terminology Criteria for Adverse Events (CTCAE version 5.0). Only adverse events that are attributed as either "possibly-", "probably-", or "definitely-" related to study drug will be assessed in the determination of tolerance. "Good" tolerance is defined as no adverse events occurring or only adverse events coded as CTCAE grades 1 and 2. "Poor" tolerance is defined as any adverse events attributed as possibly-, probably-, or definitely-related to study drug coded as CTCAE grades 3, 4, or 5.
Nested Study A1.1 Type of Short Intensive Therapy - MABS clearance from respiratory sample(s) with tolerance. | Screening (Day 0) to the End of Short Intensive Therapy (Week 6).
  To compare the microbiological clearance of MABS from respiratory samples collected at 4 weeks with good tolerability assessed at the end of short intensive therapy between the use of Inhaled Amikacin (Arm B) and the use of Intravenous Amikacin (Arm A) given during intensive phase. Definition of MABS clearance is 3 MABS negative sputum samples or ONE MABS negative Bronchoalveolar Lavage (BAL) at end of Short Intensive Therapy. "Good" tolerance is defined as no adverse events occurring or only adverse events that are attributed as either "possibly-", "probably-", or "definitely-" related to study drug coded as CTCAE grades 1 and 2.
Nested Study A1.2 - Duration of intensive therapy for patients completing short intensive treatment with ongoing positive MABS cultures collected at 4 weeks and randomised to either a further 6 weeks intensive therapy or immediate consolidation. | Screening (Day 0) to EITHER the End of Prolonged Intensive Therapy (for those allocated to Prolonged Intensive) OR Week 12 Visit (for those allocated to immediate consolidation therapy).
  To compare the microbiological clearance from samples collected at 10 weeks with good tolerability between those who are allocated to prolonged intensive therapy and those allocated to immediate consolidation following short intensive therapy.
  MABS clearance, assessed at the end of prolonged intensive therapy (for those allocated to prolonged intensive) or at 12 weeks (for those allocated to immediate consolidation) will be defined as negative MABS cultures from all 3 sputum samples or from one BAL sample collected at 10 weeks. "Good" tolerance is defined as no adverse events occurring or only adverse events that are attributed as either "possibly-", "probably-", or "definitely-" related to study drug coded as CTCAE grades 1 and 2.
Nested Study 1.3 Consolidation Therapy - The use of oral therapy only or oral therapy and inhaled amikacin for consolidation therapy. | Start of Consolidation Therapy (Date of Randomisation to Consolidation Therapy) to End of Treatment plus 4 weeks off treatment (Final Outcome Visit - Week 56 for those randomised to Immediate Consolidation or Week 62 for those in Prolonged Intensive).
  To compare the microbiological clearance with good tolerability of MABS between those allocated to consolidation therapy with oral treatment and those allocated to consolidation therapy with oral treatment and additional Inhaled Amikacin at Final Outcome.
  Definition of MABS clearance at final outcome: Negative MABS cultures from four consecutive sputum samples with one of those sputum specimens collected four weeks after the completion of consolidation therapy, or a MABS negative Bronchoalveolar Lavage (BAL) collected four weeks after completion of consolidation. "Good" tolerance is defined as no adverse events occurring or only adverse events that are attributed as either "possibly-", "probably-", or "definitely-" related to study drug coded as CTCAE grades 1 and 2.

SECONDARY OUTCOMES:
Probability of MABS clearance at Final Outcome irrespective of toxicity according to participant's treatment pathway. | Screening (Day 0); at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Probability of MABS clearance at Final Outcome irrespective of toxicity according to participant's treatment pathway. Definition of MABS clearance at final outcome: Negative MABS cultures from four consecutive sputum samples with one of those sputum specimens collected four weeks after the completion of consolidation therapy, or a MABS negative Bronchoalveolar Lavage (BAL) collected four weeks after completion of consolidation.
Safety of treatment combinations based on adverse event reporting. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Safety of treatment combinations based on the reporting of adverse events that are attributed as either "possibly-", "probably-", or "definitely-" related to study drugs.
Safety of treatments based on changes in microbiological resistance. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Safety of treatments based on changes to microbiological resistance of the MABS bacteria during the study treatment period.
Change in FEV1 z-score at Final Outcome compared with Screening in participants who do and do not clear MABS at Final Outcome. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Change in FEV1 z-score at Final Outcome compared with Screening in participants who do and do not clear MABS at Final Outcome.
Phenotype of the structural abnormalities of chest CTs and changes in chest CT scores between Screening and Final Outcome between participants who clear or do not clear MABS at Final Outcome. | Screening (Day 0); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Phenotype of the structural abnormalities of chest CTs and changes in chest CT scores between Screening and Final Outcome between participants who clear or do not clear MABS at Final Outcome.
Predictive value of structural abnormalities on Screening CT scans for sputum conversion and for progression of structural changes in relation to treatment. | Screening (Day 0); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Predictive value of structural abnormalities on Screening CT scans for sputum conversion and for progression of structural changes in relation to treatment.
Change in 6-minute walk distance (6MWD) for adult participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Change in 6-minute walk distance (6MWD) for adult participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome.
Change in HRQoL (measured using the CFQ-R) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Change in HRQoL (measured using the CFQ-R) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. CFQ-R is the Cystic Fibrosis Questionnaire Revised and will be completed by all CF participants.
Change in HRQoL (measured using the EQ-5D) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Change in HRQoL (measured using the EQ-5D) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. EQ-5D is the EuroQol 5 Dimensions and will be completed by all participants.
Change in HRQoL (measured using the SGRQ) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Change in HRQoL (measured using the SGRQ) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. SGRQ is the St George's Respiratory Questionnaire and will be completed by all non-CF participants who are 18 years and older.
Change in HRQoL (measured using the SF-36) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Change in HRQoL (measured using the SF-36) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. The SF-36 is the Short-Form 36 questionnaire and will be completed by all participants 16 years and older.
Change in HRQoL (measured using the PedsQL) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Change in HRQoL (measured using the PedsQL) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. The PedsQL is the Pediatric Quality of Life Inventory questionnaire and will be completed by participants 2 years old to 16 years old.
Change in HRQoL (measured using the CHU-9D) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Change in HRQoL (measured using the CHU-9D) for participants from Screening to Final Outcome according to treatment pathway and in participants who do and do not clear MABS at Final Outcome. CHU-9D is the Child Health Utility 9D and will be completed by all children aged 7 to 17 years of age.
Cost effectiveness of the treatment combinations (measured using the Costs Questionnaire and Linked Administrative Healthcare Utilisation Data (for applicable jurisdictions)) across intensive and consolidation phases of the trial. | Screening (Day 0); At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Cost effectiveness of the treatment combinations across intensive and consolidation phases of the trial. Cost effectiveness of the treatments will be assessed using the unvalidated "Costs Questionnaire" and where applicable and available, the linked administrative healthcare utilisation data e.g. in Australian participants.
Causes for early withdrawal from MABS-PD treatment due to reasons other than poor tolerance as defined in the primary objectives. | At End of Short Intensive Therapy (Week 6); At End of Prolonged Intensive Therapy OR at Week 12 visit; at End of Treatment plus 4 weeks off treatment (Final Outcome Visit - either Week 56 or Week 62).
  Causes for early withdrawal from MABS-PD treatment due to reasons other than poor tolerance as defined in the primary objectives.

OTHER OUTCOMES:
Participant's MABS clearance status 12 months after Final Outcome. | 12 months after End of Treatment plus 4 weeks off treatment (Final Outcome Visit).
  Participant's MABS clearance status 12 months after Final Outcome will be assessed by a 12 month follow up questionnaire that will be completed by the site investigator.

CONTACTS AND LOCATIONS:
Locations (50):
- Australia (22):
  - St George Hospital, Kogarah, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - Sunshine Coast University Hospital, Birtinya
  - Royal Prince Alfred Hospital, Camperdown
  - The Prince Charles Hospital, Chermside
  - Gold Coast University Hospital, Gold Coast
  - Greenslopes Private Hospital,, Greenslopes
  - Sir Charles Gairdiner Hospital, Nedlands
  - John Hunter Hospital, New Lambton
  - John Hunter Children's Hospital, New Lambton Heights
  - Perth Children's Hospital, Perth
  - The Alfred, Prahran
  - Sydney Children's Hospital, Randwick
  - Mater Adult Hospital, South Brisbane
  - Macquarie University Hospital, Sydney
  - The Children's Hospital at Westmead, Westmead
  - Westmead Hospital, Westmead
- Rigshospitalet, Copenhagen, Denmark
- Israel (6):
  - Soroka Medical Centre, Beer-Sheeva
  - Carmel Medical Centre, Haifa
  - Rambam Health Care Campus, Haifa
  - Hadassah Ein Kerem Hospital, Jerusalem
  - Schneider, Petah Tikva
  - Sheba Medical Centre, Ramat Gan Tel Aviv
- Erasmus MC Sophia Children's Hospital, Rotterdam, Netherlands
- Tan Tock Seng Hospital Pte Ltd, Singapore, Singapore
- Taiwan (2):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- United Kingdom (17):
  - Belfast City Hospital, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Noah's Ark Childrens Hospital for Wales, Cardiff
  - Royal Hospital for Children and Young People, Edinburgh, Edinburgh
  - Western General Hospital, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow, Glasgow
  - Alder Hey Children NHS Foundation Trust, Liverpool
  - Royal Brompton Hosptial, London
  - Royal Manchester Children's Hospital, Manchester
  - Nottingham Children's Hosptial, Nottingham
  - Queens Medical Centre, Nottingham
  - Welcome Wolfson Adult CF Centre (City Hospital Campus), Nottingham
  - University Hospital Llandough, Penarth
  - Southampton General Hospital, Southampton
  - Wythenshawe Hospital, Wythenshawe

IPD SHARING:
Plan to Share IPD: Yes
All de-identified raw data measured during the trial will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication with no end date.
Access Criteria: Data will be made available to recognised academic institutes and clinical teams upon written request with a proposal for data usage to Chief Investigator, Professor Claire Wainwright

REFERENCES:
- [Derived] Jong T, Baird T, Barr HL, Bell S, Bigirumurame T, Brady K, Burke A, Byrnes J, Caudri D, Clark JE, Coin LJM, Goh F, Grimwood K, Hicks D, Jayawardana K, Joshi S, Lee K, Qvist T, Reid D, Rice M, Roberts JA, Rogers G, Shackleton C, Sly PD, Smyth AR, Stevens L, Stockwell R, Tarique A, Taylor S, Thomson R, Tiddens HAWM, Wang XF, Wason J, Wainwright C. Finding the optimal regimen for Mycobacteroides abscessus treatment (FORMaT) in people with Mycobacteroides abscessus pulmonary disease: a multicentre, randomised, multi-arm, adaptive platform trial. BMJ Open. 2025 Sep 21;15(9):e096188. doi: 10.1136/bmjopen-2024-096188. PMID 40976660

DOCUMENTS (1):
  • Study Protocol (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT04310930/Prot_004.pdf